CLINICAL TRIAL: NCT00661401
Title: Serum IgG Antibody to Streptococcus Pneumoniae, Haemophilus Influenzae Type b and Tetanus Toxoid in Patients With Primary Antibody Deficiencies Treated With Subcutaneous Immunoglobulin Infusions
Brief Title: Specific IgG Antibody in Patients With Primary Antibody Deficiencies Treated With Subcutaneous Immunoglobulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Albertina da Rosa Borges Pizzamiglio, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 310570; 315970
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Common Variable Immunodeficiency; Agammaglobulinemia
Keywords: gammaglobulin; subcutaneous infusion; specific antibodies; primary antibody deficiency
MeSH Terms: conditions — Common Variable Immunodeficiency; Agammaglobulinemia; Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: gammaglobulin — They were administered a polyvalent, pasteurized liquid immune globulin subcutaneously (human 16% Beriglobin ®, Germany) with doses ranging from 57 to 132 mg/kg/week in order to maintain the same dosage they received by intravenous route monthly previous to this protocol. After a wash-out period (15 weeks) of the subcutaneous immunoglobulin administration, blood was collected every 4 weeks immediately before infusions. The infusions were administered using battery-powered ambulatory syringe drivers together with 10 or 20 ml syringe and infusions sets according to a pre-defined protocol (Gardulf et al, 2006).
  Other Names: Beriglobin 17540311E

SUMMARY:
Objective: Measure serum IgG antibody to Streptococcus pneumoniae serotypes 1, 3, 5, 6B, 9V e 14, Haemophilus influenzae type b and tetanus toxoid in patients with primary antibody deficiencies who were treated with subcutaneous immunoglobulin infusions.

DETAILED DESCRIPTION:
Therapy with polyvalent immunoglobulin (Ig) has been established as the standard therapy for antibody deficiencies for several decades now. Although subcutaneous infusions were originally proposed as an alternative to intramuscular injections, more recently, this method has been proven as a safe and convenient method for providing immunoglobulin levels in adults and children. Subcutaneous administration of immunoglobulins has some clinical advantages over intravenous immunoglobulin infusions (IVIG) , including a more benign side effect profile, better sustained levels of IgG in the blood and reduced cost. An additional benefit is an improvement in the quality of life, which is in part secondary to the feasibility of the patients to administer it themselves at home. The most common infections in primary antibody deficiency patients involves encapsulated bacteria, mainly Streptococcus pneumoniae and Haemophilus influenzae type b. The aim of this study is to verify if patients with antibody deficiency receiving subcutaneous immunoglobulin (SCIG) infusions keep protective antibody levels to Streptococcus pneumoniae, Haemophilus influenzae type b (Hib) and tetanus toxoid.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of a primary immunodeficiency disease with hypo-or agammaglobulinemia
* diagnosis performed according to the WHO definitions
* already been treated with Intravenous immunoglobulin or subcutaneous immunoglobulin for at least 6 months prior to enrollment into this study
* documented IgG trough levels (at least two values), type of used IgG preparation, dosage and dosage interval over a period of 6 months prior to enrollment into this study

Exclusion Criteria:

* history of hypersensitivity to the study medication or to drugs with similar chemical structures
* hypersensitivity to IgA
* subjects currently requiring <400 or > 600 mg/kg/b.w. immunoglobulin per month
* subjects whose dosage intervals for IV Ig are < 3 weeks
* know pregnancy or positive pregnancy test
* nursing mothers
* childbearing potential, if an acceptable birth control is not practiced
* history of chronic or persisting renal insufficiency (serum creatinine above upper limit of normal)
* history of chronic or persisting hepatic insufficiency (ALT> 2 times the upper limit of normal)
* risk of developing acute renal failure (Diabetes mellitus, volume depletion, sepsis, paraproteinemia)
* any symptomatic heart disease requiring treatment (NYHA class II or above)
* history of seizure disorder
* history or risk for occlusive vascular disease
* indication of active hepatitis A, B, or C at screening (HAV-PCR, HBV-PCR, or HCV-PCR positive)
* detection of HIV-1 PCR positive
* likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* progressive fatal disease/life expectancy of less than 12 months
* history of drug or alcohol abuse
* pathological mental condition rendering the subject unable to understand, scope and possible consequences of the study and/or evidence of an uncooperative attitude
* treatment with nephrotoxic drugs during the last 3 weeks
* treatment with any other investigational drug in the last 3 months before study entry or likelihood of treatment with another investigational grug during the study period
* evidence of uncooperative attitude
* vaccination against hepatitis B within 3 months before enrollment into the study
* former participation in this trial

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2002-01; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Specific IgG levels were measured using ELISA. Adequate response was arbitrarily defined as equal to or higher than 1.3 mg/L to pneumococci (Sorensen RU et al 1998), 1.0 mg/L to Hib (Takano AO 1997) and 0.1 IU/mL to tetanus toxoid (Kayhtyh et al 1983). | Samples from patients blood was collected every 4 weeks on 7 different occasions immediately before infusions.All patients were treated with subcutaneous immunoglobulin for 43 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz T Costa Carvalho, md PhD, Study Director — Federal University of São Paulo; Charles K Naspitz, md MSc, Study Chair — Federal University of São Paulo; Albertina RB Pizzamiglio, md MSc, Principal Investigator — Federal University of São Paulo; Aparecida T Nagao-Dias, Study Director — Federal University of Ceará
Locations (1):
- Division of Allergy, Clinical Immunology and Rheumatology, Department of Pediatrics, Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Gardulf A, Nicolay U, Asensio O, Bernatowska E, Bock A, Carvalho BC, Granert C, Haag S, Hernandez D, Kiessling P, Kus J, Pons J, Niehues T, Schmidt S, Schulze I, Borte M. Rapid subcutaneous IgG replacement therapy is effective and safe in children and adults with primary immunodeficiencies--a prospective, multi-national study. J Clin Immunol. 2006 Mar;26(2):177-85. doi: 10.1007/s10875-006-9002-x. Epub 2006 Apr 26. PMID 16758340
- [Background] Sorensen RU, Leiva LE, Javier FC 3rd, Sacerdote DM, Bradford N, Butler B, Giangrosso PA, Moore C. Influence of age on the response to Streptococcus pneumoniae vaccine in patients with recurrent infections and normal immunoglobulin concentrations. J Allergy Clin Immunol. 1998 Aug;102(2):215-21. doi: 10.1016/s0091-6749(98)70089-2. PMID 9723664
- [Background] Kayhty H, Peltola H, Karanko V, Makela PH. The protective level of serum antibodies to the capsular polysaccharide of Haemophilus influenzae type b. J Infect Dis. 1983 Jun;147(6):1100. doi: 10.1093/infdis/147.6.1100. No abstract available. PMID 6602191
- [Background] Pichichero ME, Anderson EL, Rennels MB, Edwards KM, England JA. Fifth vaccination with dipthteria, tetanus and acellular pertussis is beneficial in four- to six-year-olds. Pediatr Infect Dis J. 2001 Apr;20(4):427-33. doi: 10.1097/00006454-200104000-00011. PMID 11332669